CLINICAL TRIAL: NCT03045666
Title: The Impact of Macitentan Therapy and Rehabilitation Program on Peak Oxygen Consumption in Patients With Severe Pulmonary Arterial Hypertension
Brief Title: Impact of Rehabilitation Program on PAH Patients Treated With Macitentan.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SOR-026116-CTIL
Record Dates: First submitted 2017-02-05; First posted 2017-02-07 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Resistance Training; Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients stable on Macitentan therapy will exercise twice a week for 12 weeks, supervised by physiotherapists. The exercise program includes aerobic and strength exercises, at 2-3 minutes intervals.
  Interventions: Other: Exercise program
- Control Group (No Intervention): Patients stable on Macitentan therapy that will continue to receive it, without exercise.

INTERVENTIONS:
Other: Exercise program — patients who are stable on Macitentan therapy (received in both groups before enrollment) and will exercise at a pulmonary rehabilitation program twice a week for 12 weeks
  Other Names: Rehabilitation program
  Arms: Intervention group

SUMMARY:
48 patients, over the age of 18, with pulmonary arterial hypertension (PAH) classified as WHO III-IV, that are all stable under Macitentan therapy ( medication for treating PAH patients), will be recruited to the study through the pulmonary hypertension (PH) clinic at Soroka Medical Center. The patients will be randomly divided into an intervention group, which will exercise twice a week for 12 weeks, supervised by physiotherapists, and a control group, which will only receive the medication. Tests will be performed before the beginning of the intervention program, 6 weeks after it has begun, at the end of the 12 week program, and 3 months after finishing the program.

DETAILED DESCRIPTION:
48 patients, over the age of 18, with PAH classified as WHO III-IV, that are all stable under Macitentan therapy, will be recruited to the study through the PH clinic at Soroka Medical Center. The patients will be randomly divided into intervention and control groups.

The intervention group will exercise in a pulmonary rehabilitation program twice a week, for 12 weeks. The exercise protocol will include circuit training, with 2-3 minutes exercise intervals, including aerobic and strength training, and will be supervised by physiotherapists. The control group will continue to receive their usual Macitentan treatment.

All study participants will undergo tests before the beginning of the intervention program, 6 weeks after it has begun, at the end of the 12 week program, and 3 months after finishing the program. The tests will include a cardio-pulmonary exercise test, 6 minute walk distance measurement, WHO functional class evaluation, levels of Brain natriuretic peptide (BNP), EMPHASIS10 questionnaire (emPHasis-10 questionnaire is a short questionnaire for assessing Health Related Quality of Life in pulmonary arterial hypertension), Short Form-36 (SF-36) quality of life questionnaire and echocardiography.

Once data collection is completed, two way ANOVA repeated measures will be used to assess the changes in outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. PAH patients group 1
2. Patients Age > 18 years,
3. Patients with WHO III
4. Patients on Macitentan treatment who are stable on disease-targeted medication for at least 2 months prior to inclusion.

Exclusion Criteria:

1. Patients with other significant comorbidity such as Pulmonary veno-occlusive disease (PVOD) or pulmonary capillary haemangiomatosis, Malignancy, Recent myocardial infarction in the last 2 weeks.
2. Patients on other PAH specific medications treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-04-15 (Estimated); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Cardio-pulmonary exercise test- measurements of VO2 , anaerobic threshold, respiratory exchange ratio, O2 pulse, ventilatory reserve, heart rate, End tidal CO2 and O2, work rate, ventilation (VE), VCO2 during exercise test | 0-24 weeks
  Physiological response to exercise

SECONDARY OUTCOMES:
Echocardiography: dimensions and pressure of left and right ventricles, cardiac output, pulmonary arterial pressure (systolic, diastolic and mean), pulmonary capillary wedge pressure | 0-12 weeks
  Cardiac function
EMPHASIS10 questionnaire | 0-24 weeks
  Disease specific quality of life questionnaire
SF-36 questionnaire | 0-24 weeks
  Quality of life questionnaire
N-terminal prohormone brain natriuretic peptide (NT-proBNP) | 0-12 weeks
  high levels of NT-proBNP can indicate heart failure
Functional class evaluation | 0-24 weeks
  Functional class as classified by the world health organization (WHO)
6 minute walk distance | 0-24 weeks
  Functional capacity assesment by 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Avital Abriel Keren, Principal Investigator — Soroka University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided